CLINICAL TRIAL: NCT03050112
Title: Long-term Quality of Life of Patients With a Congenital Heart Disease, Treated by Surgery in Adulthood at the Brugmann Hospital.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUB-QOL cardiopathy
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Congenital Heart Disease
Keywords: MacNew questionnaire; Quality of life
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Congenital cardiopathy (Experimental): Patients having had surgery in adulthood for a congenital heart disease, at the Brugmann University Hospital. The group consists in patients aged 16 years or older, having had surgery between 01/01/1998 and 31/12/2015.
  Interventions: Other: MacNew questionnaire

INTERVENTIONS:
Other: MacNew questionnaire — Patients will be asked to fill in the MacNew questionnaire on quality of life (phone contact).

SUMMARY:
Adults with a congenital heart disease, having undergone a surgical intervention or a re-do surgery in adulthood, are a growing group of subjects in the general population. This increase is explained by improved medical and surgical techniques, with a better survival rate as outcome.

There is nowadays a growing interest in the quality of life of this group of subjects. However, studies give contradictory results. This can be explained on one hand by the vast majority of pathologies within this population, and on the other hand by the absence of a cardio-specific tool for quality of life measurement.

The MacNew questionnaire is cardio-specific. It allows an evaluation of the quality of life based on the exploration of three domains: physical, emotional and social.

The aim of this study is:

* to evaluate the quality of life of these patients, by using the MacNew questionnaire
* to explore the needs in terms of prevention, treatment and multi-disciplinary follow-up
* to assess the mortality within this group of patients.

ELIGIBILITY:
Inclusion Criteria:

Patients having had surgery in adulthood for a congenital heart disease, at the Brugmann University Hospital. The group consists in patients aged 16 years or older, having had surgery between 01/01/1998 and 31/12/2015

Exclusion Criteria:

None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
MacNew questionnaire | 30 minutes
  Quality of life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Halit Ozel, Principal Investigator — CHU Brugmann; Pierre Wauthy, MD, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wauthy P, Massaut J, Sanoussi A, Demanet H, Morissens M, Damry N, Dessy H, Malekzadeh-Milani SG, Deuvaert FE. Ten-year experience with surgical treatment of adults with congenital cardiac disease. Cardiol Young. 2011 Feb;21(1):39-45. doi: 10.1017/S1047951110001332. Epub 2010 Oct 6. PMID 20923595
- [Background] Lane DA, Lip GY, Millane TA. Quality of life in adults with congenital heart disease. Heart. 2002 Jul;88(1):71-5. doi: 10.1136/heart.88.1.71. PMID 12067950
- [Background] Immer FF, Althaus SM, Berdat PA, Saner H, Carrel TP. Quality of life and specific problems after cardiac surgery in adolescents and adults with congenital heart diseases. Eur J Cardiovasc Prev Rehabil. 2005 Apr;12(2):138-43. doi: 10.1097/01.hjr.0000159318.62466.dc. PMID 15785299
- [Background] Fteropoulli T, Stygall J, Cullen S, Deanfield J, Newman SP. Quality of life of adult congenital heart disease patients: a systematic review of the literature. Cardiol Young. 2013 Aug;23(4):473-85. doi: 10.1017/S1047951112002351. Epub 2013 Feb 6. PMID 23388149
- [Background] Apers S, Luyckx K, Moons P. Quality of life in adult congenital heart disease: what do we already know and what do we still need to know? Curr Cardiol Rep. 2013 Oct;15(10):407. doi: 10.1007/s11886-013-0407-x. PMID 23955787
- [Background] Hofer S, Lim L, Guyatt G, Oldridge N. The MacNew Heart Disease health-related quality of life instrument: a summary. Health Qual Life Outcomes. 2004 Jan 8;2:3. doi: 10.1186/1477-7525-2-3. PMID 14713315
- [Background] Pavy B, Iliou MC, Hofer S, Verges-Patois B, Corone S, Aeberhard P, Curnier D, Henry J, Ponchon-Weess A, Oldridge N. Validation of the French version of the MacNew heart disease health-related quality of life questionnaire. Arch Cardiovasc Dis. 2015 Feb;108(2):107-17. doi: 10.1016/j.acvd.2014.09.006. Epub 2014 Nov 12. PMID 25453715
- [Background] Dixon T, Lim LL, Oldridge NB. The MacNew heart disease health-related quality of life instrument: reference data for users. Qual Life Res. 2002 Mar;11(2):173-83. doi: 10.1023/a:1015005109731. PMID 12018740